CLINICAL TRIAL: NCT03279510
Title: Hearing Aids and the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2396-P
Record Dates: First submitted 2017-08-23; First posted 2017-09-12 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Hearing Loss
Keywords: auditory perception; hearing
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hearing aids (Experimental): All study participants will be fit with hearing aids.
  Interventions: Device: hearing aids

INTERVENTIONS:
Device: hearing aids — Subjects are fit with hearing aids.

SUMMARY:
Hearing aids are being fit on inexperienced hearing aid users and the short-term and long-term effects are measured. This research aims to improve understanding of the individual factors that contribute to receiving benefit from hearing aids and lead to more individualized treatment of hearing loss.

DETAILED DESCRIPTION:
Hearing aids are used to improve audibility for patients with hearing loss and improve speech perception. In addition to these immediate benefits, amplification has the potential to have long-term effects on higher level auditory processing abilities, such as cognition or other abilities required for complex listening tasks. These long-term acclimatization effects are not well understood and merit further behavioral and physiological examination. Hearing aids will be fit on inexperienced hearing aid users and outcome measures will be used to determine immediate and long-term effects of hearing aids. This research may provide a more detailed view of individual differences that contribute to receiving benefit from a hearing aid and may lead to more individualized treatment of hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Bilateral, mild to moderately severe hearing loss
* Inexperienced hearing aid users

Exclusion Criteria:

* Subject deciding that they do not wish to wear hearing aids as necessitated per study protocol
* Audiometric thresholds that suggest research stimuli would not be audible
* Conductive hearing loss and/or other significant ear or hearing problems
* Non-native English speakers
* Conditions or circumstances that would preclude a participant from wearing hearing aids consistently or finishing the study
* An inability to perform or complete the experimental tasks

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Evoked potential latency | Approximately 1 year
  Latency will be measured in milliseconds
Evoked potential amplitude | Approximately 1 year
  Amplitude will be measured in microvolts
Frequency following response magnitude | Approximately 1 year
  Magnitude of response measured in nanovolts
Frequency following response timing | Approximately 1 year
  Timing measured by cross-correlation between stimulus and response
Ongoing electroencephalography power | Approximately 1 year
  EEG power as a function of frequency recorded during words-in-noise measure
Montreal Cognitive Assessment score | Approximately 1 year
  Assessment score from 1 to 30
Reading Span | Approximately 1 year
  Percent correct recall on working memory task
Hearing aid usage | Approximately 1 year
  Data logging from the hearing aid will provide usage in hours per day
Word-in-noise perception testing | Approximately 1 year
  Signal-to-noise ratio at which participant correctly understands 50% of speech in noise using WIN test
Listening invested/required effort | Approximately 1 year
  Participants' rating of the effort required (0-9) and invested (0-9) for listening task
Working memory testing | Approximately 1 year
  Performance on auditory working memory task
Glasgow Hearing Aid Benefit Profile (GHABP) | Approximately 1 year
  Participants rating on five-point scale their perceived initial (i.e., unaided) hearing disability, initial handicap, aided benefit, aided handicap, HA use and HA satisfaction in four listening situations

CONTACTS AND LOCATIONS:
Overall Officials: Curtis J. Billings, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No